CLINICAL TRIAL: NCT05073835
Title: BARI-STEP:A Double-blinded, Randomised, Placebo-controlled Trial of Semaglutide 2.4 mg in Patients With Poor Weight-loss Following Bariatric Surgery.
Brief Title: Semaglutide 2.4 mg in Patients With Poor Weight-loss
Acronym: BARI-STEP
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University College, London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 142522
Record Dates: First submitted 2021-09-15; First posted 2021-10-12 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Obesity; Diabetes; Metabolic Syndrome
Keywords: obesity; diabetes; semaglutide
MeSH Terms: conditions — Obesity; Diabetes Mellitus; Metabolic Syndrome | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: Phase 3b, double-blinded, randomised, parallel group trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: double blinded: both participants and study doctors will be blind to group allocation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Semaglutide 2.4mg/week subcutaneous injection for 68 weeks. The treatment includes an initial 16-week escalation phase followed by 52 weeks of treatment at study dose, i.e., 2.4mg/week.
  Interventions: Drug: Semaglutide 3 mg
- Control (Placebo Comparator): Placebo administration, once weekly, subcutaneous injection.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Semaglutide 3 mg — Semaglutide 2.4 mg/week, subcutaneous injection. Treatment dose: 16 weeks of dose escalation + 52 weeks of study dose (i.e., 2.4 mg/week).
  Arms: Intervention
Drug: Placebo — Placebo
  Arms: Control

SUMMARY:
A double-blinded, randomised, placebo-controlled trial of semaglutide 3.0 mg/ml in patients with poor weight-loss following bariatric surgery. The primary aim of this trial is to determine whether, and the extent to which, 68 weeks of subcutaneous semaglutide 3.0 mg/ml causes greater percentage weight loss (%WL), reduction in adiposity, improvement in metabolic and inflammatory indices and health-related quality of life (HRQoL) than placebo, in patients with poor weight loss following gastric bypass or sleeve gastrectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Patients, ≥1 year primary GB or primary SG, with poor weight-loss (<20% WL) that is not caused by either a surgical or psychological problem.
2. Adults, 18-65 years inclusive.
3. Females of childbearing potential and female partners of male participants must be willing to use highly effective method of contraception (hormonal or barrier method of birth control; abstinence) (Appendix 2) from the time consent is signed until 2 months after treatment discontinuation.
4. Females of childbearing potential must have a negative pregnancy test within 7 days prior to randomisation. NOTE: Subjects are considered not of child bearing potential if they are surgically sterile (i.e. they have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are postmenopausal.
5. A self-reported ≤5 % variation in body weight over preceding 3 months.
6. Fluent in English and able to understand and complete questionnaires.
7. Participants capable to provide written informed consent and comply with the trial protocol.

Exclusion Criteria:

1. Bariatric surgical procedure other than GB and SG, or revision bariatric surgery of any operation type.
2. Personal history of type I diabetes or type II diabetes mellitus currently treated with insulin.
3. Concomitant use of GLP-1R agonist or DPPIV-inhibitors.
4. Female who is pregnant, breast-feeding, or intends to become pregnant.
5. Current participation in other clinical intervention trial.
6. History of suicidal attempt in the previous 5 years or untreated severe depression or mental health condition assessed by direct questioning.
7. Symptomatic gallstone disease
8. Uncontrolled hypertension (systolic blood pressure ≥ 160 mmHg or diastolic blood pressure ≥ 100 mmHg).
9. Renal impairment measured as glomerular infiltration rate (eGFR <15 ml/min 1.73 m2
10. Known or suspected hypersensitivity to semaglutide or any of the excipients involved in their formulation.
11. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia syndrome type 2.
12. History of malignant neoplasms within the past 5 years prior to screening. Basal and squamous cell skin cancer and any carcinoma in-situ are allowed.
13. Personal history of acute pancreatitis 180 days before screening or chronic pancreatitis.
14. Uncontrolled thyroid disease.
15. History of stroke, unstable angina, acute coronary syndrome, congestive heart failure New York Heart Association class III-IV within the preceding 12 months.
16. Untreated clinically significant arrhythmias.
17. Diabetic gastroparesis.
18. Concomitant usage of medications that cause weight gain or weight loss.
19. Known or suspected abuse of alcohol or recreational drugs.
20. Severe hepatic impairment diagnosed via liver function blood tests and clinical evaluation
21. Any additional factor, which in the investigator's opinion, might jeopardise the subject's safety or compliance with the trial protocol.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-03 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Weight loss | 68 weeks
  Percentage of total weight loss

SECONDARY OUTCOMES:
body weight reduction ≥10% | 68 weeks
  To compare the percentage of participants receiving subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo who after 68 weeks achieve a body weight reduction ≥10%
body weight reduction ≥15% | 68 weeks
  To compare the percentage of participants receiving subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo who after 68 weeks achieve a body weight reduction ≥15%
body weight reduction ≥20% | 68 weeks
  To compare the percentage of participants receiving subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo who after 68 weeks achieve a body weight reduction ≥20%
Change in circulating HbA1c levels | 68 weeks
  The effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon HbA1c
Change in circulating HbA1c levels in participants with pre-diabetes at baseline | 68 weeks
  The effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon HbA1c in participants with pre-diabetes at baseline
Change in circulating HbA1c levels in participants with T2D at baseline | 68 weeks
  The effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon HbA1c in participants with diabetes at baseline
Systolic and diastolic BP | 68 weeks
  The effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon BP
Systolic and diastolic BP in participants with pre-existing hypertension | 68 weeks
  The effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon BP in participants with pre-existing hypertension
pharmacological agents required for the management of hypertension | 68 weeks
  The number of pharmacological agents required for the management of hypertension in participants with pre-existing hypertension
Change in circulating lipids | 68 weeks
  To compare the effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon circulating lipids
Change in circulating HsCRP and inflammatory cytokines | 68 weeks
  To compare the effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon inflammatory markers
Changes in food craving scores assessed through power of food questionnaire | 68 weeks
  To compare the effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon food cravings
Changes in HRQoL | 68 weeks
  To compare the effect of 68 weeks of subcutaneous semaglutide 3.0 mg/ml at a dose of 2.4mg per week versus placebo administration upon HRQoL
GLP-1 levels | 68 weeks
  To investigate the relationship between fasted and meal-stimulated active GLP-1 levels at baseline and %WL at 68 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Janine Makaronids, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided